CLINICAL TRIAL: NCT03982511
Title: Improving Parent-Child Interactions to Prevent Child Obesity in Early Childhood
Brief Title: Improving Parent-Child Interactions to Enhance Child Health
Acronym: PCIT-Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Michigan University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F63376; R21HD093944 (NIH)
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-02

CONDITIONS: Child Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Parent-child dyads will be randomly assigned to PCIT-Health or a waitlist control.
Who Masked: Outcomes Assessor
Masking Description: Behavioral observation coders are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCIT-Health (Experimental): Participants assigned to the PCIT-Health arm will receive the intervention.
  Interventions: Behavioral: PCIT-Health
- Wait list control (No Intervention): Participants in the wait list control will receive an invitation to participate in the intervention 10 months after baseline data collection.

INTERVENTIONS:
Behavioral: PCIT-Health — PCIT-Health (also known as Parents Active in Their Children's Health; PATCH) is an adaptation of Parent-Child Interaction Therapy. PCIT-Health targets (1) the parent-child relationship and (2) parenting efficacy both in general contexts (child play time and clean up time) and specifically in the context of obesity risk-related behaviors (child feeding, family mealtime, and child screen time).
  Other Names: PATCH Program
  Arms: PCIT-Health

SUMMARY:
Childhood obesity is a formidable public health issue in the United States, disproportionately affecting children from lower socioeconomic status households. Onset of obesity predicts cardiometabolic risks and other health problems in adolescence and into adulthood; thus, effective and early prevention is critical. Healthy parenting may play a pivotal role in preventing early childhood obesity. Warm, responsive, and consistent parenting is associated with the development of child self-regulation as well as healthy eating and physical activity practices, and thus may be protective against obesity risk. Targeting the parent-child relationship may be especially important when facilitating behavior change in parents who have ongoing stressors (e.g., low-income families). The proposed study aims to test an adaptation of Parent-Child Interaction Therapy (PCIT), an innovative parent management program that improves the parent-child relationship and enhances general parenting skills through the use of therapeutic in vivo coaching. Our adapted version, PCIT-Health, is a selective-prevention intervention that includes content specific to improving parent-child interactions and parenting in obesity-salient contexts, such as mealtime and child screen time. This project will elucidate novel approaches to, and novel targets of, early childhood obesity prevention and will provide data critical to test PCIT-Health in a large-scale randomized controlled trial. Parent-child dyads will be randomly assigned to PCIT-Health or a waitlist control in order to accomplish the following aims: AIM 1: To assess the acceptability and feasibility of the PCIT-Health delivery and assessment methods in low-income parents of overweight young children ages 3 to 6 years. AIM 2: To test the preliminary efficacy and estimate the effect size of PCIT-Health on changes in child BMI z-score (primary outcome) from baseline to (1) intervention completion and (2) 6-month post-intervention. AIM 3: To explore the effect of PCIT-Health on the following secondary outcomes: (1) parent-child relationship quality, (2) parent behavior management skills, (3) child self-regulation, (4) child eating behaviors, (5) child physical activity, and (6) child screen media use.

ELIGIBILITY:
Inclusion Criteria:

* child BMI > 5th percentile
* child born at 37+ weeks gestation, with no significant neo- or perinatal complications.

Exclusion Criteria:

* Child is experiencing clinical levels of behavior problems
* History of food allergies or medical problems or medications affecting appetite or weight
* Non-fluency in English
* Significant child or parent developmental delay
* Child currently in State custody
* Family currently involved with Child Protective Services
* Caregiver is receiving or has plans to receive other behavioral parenting interventions

Ages: 30 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Domoff, PhD, Principal Investigator — Central Michigan University
Locations (1):
- Center for Children, Families, and Communities, Mount Pleasant, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment (providing consent), but before assignment, two families declined to continue participating in the study. (n = 4).
Groups:
- PCIT-Health: Participants assigned to the PCIT-Health arm will receive the intervention.
  PCIT-Health: PCIT-Health (also known as Parents Active in Their Children's Health; PATCH) is an adaptation of Parent-Child Interaction Therapy. PCIT-Health targets (1) the parent-child relationship and (2) parenting efficacy both in general contexts (child play time and clean up time) and specifically in the context of obesity risk-related behaviors (child feeding, family mealtime, and child screen time). Due to the pandemic, telehealth PCIT-Health was provided to most of the participants.
Period: Overall Study
Arm/Group | PCIT-Health | Wait List Control
Started | 41 (27 caregivers and 14 children (from 14 families)) | 18 (11 caregivers and 7 children (from 7 families))
Completed | 30 (20 caregivers and 10 children (from 10 families)) | 15 (9 caregivers and 6 children (from 6 families))
Not Completed | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCIT-Health | Wait List Control | Total
Number analyzed (Participants) | 41 | 18 | 59
Age, Categorical [Count of Participants; unit: Participants] — Population: Separated by child and caregiver data.
  Participants
    Child: number analyzed (Participants) | 14 | 7 | 21
    Child: <=18 years | 14 | 7 | 21
    Child: Between 18 and 65 years | 0 | 0 | 0
    Child: >=65 years | 0 | 0 | 0
    Caregiver: number analyzed (Participants) | 27 | 11 | 38
    Caregiver: <=18 years | 0 | 0 | 0
    Caregiver: Between 18 and 65 years | 27 | 11 | 38
    Caregiver: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: Child age reported.
  months
    number analyzed (Participants) | 14 | 7 | 21
    (all) | 53.36 (16.06) | 50.86 (11.95) | 52.52 (14.56)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Separated by child and caregiver data.
  Participants
    Child: number analyzed (Participants) | 14 | 7 | 21
    Child: Female | 5 | 3 | 8
    Child: Male | 9 | 4 | 13
    Caregiver: number analyzed (Participants) | 27 | 11 | 38
    Caregiver: Female | 16 | 8 | 24
    Caregiver: Male | 11 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Separated by caregiver and child data.
  Participants
    Child: number analyzed (Participants) | 14 | 7 | 21
    Child: Hispanic or Latino | 1 | 2 | 3
    Child: Not Hispanic or Latino | 13 | 5 | 18
    Child: Unknown or Not Reported | 0 | 0 | 0
    Caregiver: number analyzed (Participants) | 27 | 11 | 38
    Caregiver: Hispanic or Latino | 1 | 1 | 2
    Caregiver: Not Hispanic or Latino | 26 | 10 | 36
    Caregiver: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Separated by child and caregiver data.
  Participants
    Child: number analyzed (Participants) | 14 | 7 | 21
    Child: American Indian or Alaska Native | 0 | 0 | 0
    Child: Asian | 1 | 0 | 1
    Child: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Child: Black or African American | 0 | 0 | 0
    Child: White | 12 | 5 | 17
    Child: More than one race | 1 | 2 | 3
    Child: Unknown or Not Reported | 0 | 0 | 0
    Caregiver: number analyzed (Participants) | 27 | 11 | 38
    Caregiver: American Indian or Alaska Native | 0 | 0 | 0
    Caregiver: Asian | 2 | 0 | 2
    Caregiver: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregiver: Black or African American | 2 | 0 | 2
    Caregiver: White | 23 | 11 | 34
    Caregiver: More than one race | 0 | 0 | 0
    Caregiver: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 18 | 59
Body Mass Index (BMI) z-score [Mean (Standard Deviation); unit: Z-score] — Child Body Mass Index (BMI) z-score. This z-score is a standard deviation away from the mean, based on the Centers for Disease Control and Prevention (CDC) growth charts. Higher z-scores indicate greater weight status. A Z-score of 0 equals the population mean, based on age and sex. Population: This measure was specific to child participants (child BMI z-score).
  Z-score
    number analyzed (Participants) | 14 | 7 | 21
    (all) | 0.71 (1.21) | 0.77 (0.84) | 0.73 (1.08)
BMI percentile [Mean (Standard Deviation); unit: percentile] — This measure was specific to child participants (child BMI percentile). Population: This measure was specific to child participants (child BMI percentile).
  percentile
    number analyzed (Participants) | 14 | 7 | 21
    (all) | 68.09 (30.50) | 73.94 (26.52) | 70.04 (28.70)

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Body Mass Index (BMI) Percentile
Description: Change in child BMI percentile will be calculated using standardized anthropometric measurement (height and weight) procedure
Time Frame: Pre-intervention (T1), post-intervention (T2;4 months after pre-intervention), and six-month follow-up (T3;10 months after pre-intervention)
Population: For Time 2, n = 11 for PCIT-health and n = 7 for control. For Time 3, n = 9 for PCIT-health and n = 6 for control.
Measure: Mean (Standard Error); unit: percentile
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 11 | 7
percentile
  Change in BMI percentile (T2-T1); negative values indicate decrease in BMI percentile | 3.66 (2.29) | 1.74 (3.24)
  Change in BMI percentile (T3-T1); negative values indicate decrease in BMI percentile: number analyzed (Participants) | 9 | 6
  Change in BMI percentile (T3-T1); negative values indicate decrease in BMI percentile | 1.12 (2.56) | 0.88 (3.72)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference from T2 to T1 for BMI z-score; Test type: Superiority; p = .73, ANOVA — Given that this is a pilot RCT, primary aim is to estimate effect sizes for a more fully-powered RCT. P-values will be provided in addition to effect size; Repeated measures; Mean Difference (Net) = 0.05, Standard Error of Mean 0.14 — Effect size: 0.17
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for BMI z-score from T3 to T1; Test type: Superiority; p = .98, ANOVA — Given that this is a pilot RCT (with a small n), primary aim is to estimate effect sizes for a more fully-powered RCT. Both p value and effect size will be provided; Repeated measures; Mean Difference (Net) = 0.00, Standard Error of Mean 0.18; Effect size: -0.01
Statistical Analysis 3: Comparison: PCIT-Health vs Wait List Control; Difference on difference for BMI percentile from T2 to T1; Test type: Superiority; p = 0.63, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = 1.93, Standard Error of Mean 3.97; Effect size: 0.24
Statistical Analysis 4: Comparison: PCIT-Health vs Wait List Control; Difference on difference for BMI percentile from T3 to T1; Test type: Superiority; p = 0.96, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = 0.24, Standard Error of Mean 4.51; Effect size: 0.03

2. Secondary Outcome: Child Self-regulation (Parent Report)
Description: Emotion Regulation (ER) Checklist, higher scores = greater regulation (better outcome). Mean calculation for total score, with Min=1 to Max=4
Time Frame: Pre-intervention (T1), post-intervention (T2; 4 months after pre-intervention), and six-month follow-up (T3; 10 months after pre-intervention)
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
units on a scale
  Change from T2 to T1 on ER subscale | 0.23 (0.31) | 0.03 (0.38)
  Change from T3 to T1 on ER subscale: number analyzed (Participants) | 19 | 9
  Change from T3 to T1 on ER subscale | 0.26 (0.29) | 0.26 (0.42)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for Emotion regulation subscale from T2 to T1; Test type: Superiority; p = 0.12, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = 0.20, Standard Error of Mean 0.12; Effect size: 0.79
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for emotion regulation subscale from T3 to T1; Test type: Superiority; p = 0.96, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = -0.01, Standard Error of Mean 0.14; Effect size: -0.02

3. Secondary Outcome: Child Screen Time
Description: Parent report of weekly amount of time child spends viewing/using screen media. Scores range from 0-168, with total scores reflecting sum of daily screen time across multiple types of screen media. Higher scores = more screen time.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Deviation); unit: Hours per week
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
Hours per week
  Change in weekly screen time from T2 to T1 | -5.72 (12.52) | 0.36 (18.37)
  Change in weekly screen time from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in weekly screen time from T3 to T1 | -2.92 (12.08) | -8.75 (26.62)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for child weekly screen time from T2 to T1; Test type: Superiority; p = 0.28, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = -6.08, Standard Error of Mean 5.42; Effect size: -0.41
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for child weekly screen time from T3 to T1; Test type: Superiority; p = 0.43, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = 5.83, Standard Error of Mean 7.17; Effect size: 0.42

4. Secondary Outcome: Child Physical Activity
Description: Measured by Actigraph accelerometer to assess sedentary, moderate, moderate-to-vigorous, and vigorous physical activity (MVPA)
Time Frame: as for outcome 2
Population: Smaller n due to incomplete data (not wearing actigraph for minimum number of days).
Measure: Mean (Standard Error); unit: minutes
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 10 | 6
minutes
  Change in Moderate-Vigorous Physical Activity minutes from T2 to T1 (higher scores = more activity) | 38.26 (13.78) | 2.94 (19.48)
  Change in Moderate-Vigorous Physical Activity minutes from T3 to T1 (higher scores = more activity): number analyzed (Participants) | 7 | 5
  Change in Moderate-Vigorous Physical Activity minutes from T3 to T1 (higher scores = more activity) | 32.55 (18.40) | 16.46 (24.09)
  Change in Sedentary minutes from T2 to T1 (higher scores = less activity) | -59.17 (31.46) | 5.23 (44.50)
  Change in Sedentary minutes from T3 to T1 (higher scores = less activity): number analyzed (Participants) | 7 | 5
  Change in Sedentary minutes from T3 to T1 (higher scores = less activity) | 14.59 (40.32) | -51.65 (52.79)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference score for MVPA minutes from T2 to T1; Test type: Superiority; p = 0.16, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = 35.32, Standard Error of Mean 23.86; Effect size: 0.85
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference score for MVPA minutes from T3 to T1; Test type: Superiority — Given that this is a pilot RCT (with a small n), primary aim is to estimate effect sizes for a more fully-powered RCT. Both p value and effect size will be provided; p = 0.61, ANOVA; Repeated measures; Mean Difference (Net) = 16.09, Standard Error of Mean 30.32; Effect size: 0.35
Statistical Analysis 3: Comparison: PCIT-Health vs Wait List Control; Difference on difference score for sedentary minutes from T2 to T1; Test type: Superiority; p = 0.26, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = -64.40, Standard Error of Mean 54.50; Effect size: -0.68
Statistical Analysis 4: Comparison: PCIT-Health vs Wait List Control; Difference on difference score for sedentary minutes from T3 to T1; Test type: Superiority; p = 0.34, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 66.25, Standard Error of Mean 66.43; effect size: 0.66

5. Secondary Outcome: Child Sleep (Parent Report)
Description: Measured by parent report of bedtime, wake time, and naps.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
hours
  Change in hours of sleep from T2 to T1 | -1.0 (2.25) | -0.36 (1.50)
  Change in hours of sleep from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in hours of sleep from T3 to T1 | -1.05 (2.68) | -2.44 (1.33)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for parent-reported sleep time from T2 to T1; Test type: Superiority; p = 0.41, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.64, Standard Error of Mean 0.75; effect size: -0.41
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for parent-reported sleep time from T3 to T1; Test type: Superiority; p = 0.16, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 1.39, Standard Error of Mean 0.95; effect size: 0.76

6. Secondary Outcome: Child Sleep (Via Actigraphy)
Description: Measured by Actigraph accelerometer.
Time Frame: as for outcome 2
Population: Incomplete actigraphy data due to participants wearing actigraph for fewer than minimum required days needed to calculate sleep.
Measure: Mean (Standard Error); unit: hours
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 9 | 5
hours
  Change in minutes of sleep from T2 to T1 | -10.15 (8.19) | 2.47 (12.38)
  Change in minutes of sleep from T3 to T1: number analyzed (Participants) | 7 | 5
  Change in minutes of sleep from T3 to T1 | -29.54 (10.10) | 9.29 (13.22)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for actigraphy-recorded sleep time from T2 to T1; Test type: Superiority; p = 0.42, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -12.62, Standard Error of Mean 14.84; effect size: -0.54
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for actigraphy-recorded sleep time from T3 to T1; Test type: Superiority; p = 0.04, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -38.83, Standard Error of Mean 16.61; effect size: -1.56

7. Secondary Outcome: Child Problematic Media Use
Description: Measured by the parent-report via Problematic Media Use Measure (Domoff et al., 2019). Higher scores = greater problematic media use. Total scores = mean of items; Min = 1 to Max = 5.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data. Higher scores indicate higher problematic media use.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
units on a scale
  Change in problematic media use from T2 to T1 | -0.30 (0.15) | -0.38 (0.21)
  Change in problematic media use from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in problematic media use from T3 to T1 | -0.36 (0.16) | -0.15 (0.23)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for problematic media use from T2 to T1; Test type: Superiority; p = 0.77, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 0.08, Standard Error of Mean 0.26; effect size: 0.15
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for problematic media use from T3 to T1; Test type: Superiority; p = 0.47, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.21, Standard Error of Mean 0.28; effect size: -0.38

8. Secondary Outcome: Parent-child Relationship Quality (Observed)
Description: Dyadic Parent-Child Interaction Coding System-IV (DPICS-IV) will be used. The DPICS provides a reliable measure of parent-child relationship quality (e.g., parents' child-centered skills, parent and child positive and negative physical and verbal interactions) and parent behavior management skills (e.g., use of contingent reinforcement, effective discipline, child compliance). This outcome reflects behavioral observation of parents' child-centered skills ("DO" skills) during child led play. This is a count variable that can range from 0 displayed skills (min) with no determined maximum. Higher numbers = more skills (better outcome).
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: Skills
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 19 | 11
Skills
  Change in child-centered skills from T2 to T1 | 7.65 (1.57) | 0.00 (2.12)
  Change in child-centered skills from T3 to T1: number analyzed (Participants) | 17 | 9
  Change in child-centered skills from T3 to T1 | 6.35 (1.99) | -0.11 (2.73)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for child-centered skills from T2 to T1; Test type: Superiority; p = 0.005, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 9.11, Standard Error of Mean 2.76; effect size: 1.65
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for child-centered skills from T3 to T1; Test type: Superiority; p = 0.05, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 8.22, Standard Error of Mean 3.81; effect size: 1.20

9. Secondary Outcome: Parent-child Relationship Quality (Parent Report)
Description: Scores on the Parent-child Dysfunctional Interaction (PCDI) subscale of the Parenting Stress Index will be used as the parent-report of parent-child relationship quality. Values range from 12 to 60, with higher scores indicating greater dysfunction in (poorer quality of) the parent-child relationship.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
score on a scale
  Change in PCDI from T2 to T1 | -9.59 (4.00) | 7.64 (5.66)
  Change in PCDI from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in PCDI from T3 to T1 | -13.21 (3.63) | 6.22 (5.27)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for PCDI scores from T2 to T1; Test type: Superiority; p = 0.02, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -17.23, Standard Error of Mean 6.93; effect size: -1.21
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for PCDI scores from T3 to T1; Test type: Superiority; p = 0.008, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -19.43, Standard Error of Mean 6.40; effect size: -1.57

10. Secondary Outcome: Pressure to Eat (Parent-report)
Description: Scores on the Child Feeding Questionnaire (CFQ)- Pressure to Eat subscale will be calculated. This subscale score is a mean, with minimum of 1 and maximum of 5 (higher scores = more pressure to eat, a worse outcome).
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
score on a scale
  Change in pressure to eat scores from T2 to T1 | -0.84 (0.21) | -0.59 (0.29)
  Change in pressure to eat scores from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in pressure to eat scores from T3 to T1 | -0.59 (0.21) | -0.58 (0.31)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for pressure to eat scores from T2 to T1; Test type: Superiority; p = 0.50, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = -0.25, Standard Error of Mean 0.36; effect size: -0.34
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for pressure to eat scores from T3 to T1; Test type: Superiority; p = 0.98, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.01, Standard Error of Mean 0.37; effect size: -0.01

11. Secondary Outcome: Restriction (Parent-report)
Description: Scores on the Child Feeding Questionnaire (CFQ)-Restriction subscale will be calculated. A mean is calculated for this subscale (min = 1 to max = 5). Higher scores = greater restriction of food (poorer outcome).
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
score on a scale
  Change in Restriction scores from T2 to T1 | -0.71 (0.18) | -0.25 (0.26)
  Change in Restriction scores from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in Restriction scores from T3 to T1 | -0.88 (0.20) | -0.53 (0.29)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for restrictive feeding scores from T2 to T1; Test type: Superiority; p = 0.17, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.46, Standard Error of Mean 0.32; effect size: -0.70
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for restrictive feeding scores from T3 to T1; Test type: Superiority; p = 0.34, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.35, Standard Error of Mean 0.35; effect size: -0.51

12. Secondary Outcome: Emotional Feeding (Parent-report)
Description: Child Feeding Questionnaire (CFQ)- Emotional Feeding subscale will be calculated with a mean of responses to items. Min = 1 to max = 5. Higher scores reflect worse outcome.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
score on a scale
  Change in emotional feeding from T2 to T1 | -0.19 (0.13) | -0.16 (0.19)
  Change in emotional feeding from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in emotional feeding from T3 to T1 | -0.37 (0.12) | -0.20 (0.18)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for emotional feeding scores from T2 to T1; Test type: Superiority; p = 0.91, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.03, Standard Error of Mean 0.23; effect size: -0.06
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for emotional feeding scores from T3 to T1; Test type: Superiority; p = 0.45, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.17, Standard Error of Mean 0.22; effect size: -0.40

13. Secondary Outcome: Instrumental Feeding (Parent-report)
Description: Scores on the Parental Feeding Questionnaire (PFQ)- Instrumental Feeding subscale will be calculated. Mean calculation of responses, with scores ranging from 1 (min) to 5 (max). Higher scores reflect poorer outcome.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
score on a scale
  Change in instrumental feeding from T2 to T1 | -0.74 (0.12) | -0.27 (0.16)
  Change in instrumental feeding from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in instrumental feeding from T3 to T1 | -0.91 (0.13) | -0.36 (0.19)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for instrumental feeding scores from T2 to T1; Test type: Superiority; p = 0.03, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.47, Standard Error of Mean 0.20; effect size: -1.12
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for instrumental feeding scores from T3 to T1; Test type: Superiority; p = 0.03, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.55, Standard Error of Mean 0.23; effect size: -1.25

14. Secondary Outcome: Active Mediation of Television (Parent-report)
Description: Scores on the Instructive Mediation subscale of the Parental Mediation Scale (Valkenburg et al., 1999) will be calculated via sum score of 5 items. Min = 5, max = 20, higher scores = better outcome.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
score on a scale
  Change in active mediation from T2 to T1 | 2.86 (0.61) | 0.64 (0.86)
  Change in active mediation from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in active mediation from T3 to T1 | 2.95 (0.84) | 0.44 (1.21)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for active mediation from T2 to T1; Test type: Superiority; p = 0.05, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 2.23, Standard Error of Mean 1.06; effect size: 1.02
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for active mediation scores from T3 to T1; Test type: Superiority; p = 0.11, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 2.50, Standard Error of Mean 1.47; effect size: 0.88

15. Secondary Outcome: Restrictive Mediation of Television (Parent-report)
Description: Scores on the Restrictive Mediation subscale of the Parental Mediation Scale (Valkenburg et al., 1999) will be calculated via sum score of 5 items. Min = 5, max = 20, higher scores = better outcome.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
score on a scale
  Change in restrictive mediation from T2 to T1 | 2.36 (0.57) | -1.27 (0.81)
  Change in restrictive mediation from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in restrictive mediation from T3 to T1 | 1.53 (0.61) | 0.22 (0.89)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for restrictive mediation scores from T2 to T1; Test type: Superiority; p = 0.002, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 3.64, Standard Error of Mean 1.00; effect size: 1.77
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for restrictive mediation scores from T3 to T1; Test type: Superiority; p = 0.24, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 1.30, Standard Error of Mean 1.08; effect size: 0.63

16. Secondary Outcome: Social Coviewing of Television (Parent-report)
Description: Scores on the Social Coviewing subscale of the Parental Mediation Scale (Valkenburg et al., 1999) will be calculated via sum score of 5 items. Min = 5, max = 20, higher scores = better outcome.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
score on a scale
  Change in social coviewing from T2 to T1 | 1.14 (0.61) | 0.45 (0.86)
  Change in social coviewing from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in social coviewing from T3 to T1 | 1.11 (0.63) | 0.78 (0.91)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for social coviewing from T2 to T1; Test type: Superiority; p = 0.53, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 0.68, Standard Error of Mean 1.05; effect size: 0.31
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for social coviewing from T3 to T1; Test type: Superiority; p = 0.77, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 0.33, Standard Error of Mean 1.10; effect size: 0.15

17. Secondary Outcome: Location/Quantity of Screen Media in the Home (Parent-report)
Description: Parents will report on the location/quantity of screen media in home and child's bedroom.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: number of screens
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 19
number of screens
  Change in number of screens in the home from T2 to T1 | 0.32 (0.89) | 0.18 (1.18)
  Change in number of screens in the home from T3 to T1 | 0.49 (0.94) | -0.39 (1.30)
  Change in number of screens in the child's bedroom from T2 to T1 | -0.21 (0.22) | 0.19 (0.30)
  Change in number of screens in the child's bedroom from T3 to T1 | -0.58 (0.22) | 0.33 (0.32)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for number of screens in the home from T2 to T1; Test type: Superiority; p = 0.91, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 0.14, Standard Error of Mean 1.23; effect size: 0.04
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for number of screens in the home from T3 to T1; Test type: Superiority; p = 0.64, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 0.65, Standard Error of Mean 1.36; effect size: 0.17
Statistical Analysis 3: Comparison: PCIT-Health vs Wait List Control; Difference on difference for number of screens in child bedroom from T2 to T1; Test type: Superiority; p = 0.31, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.36, Standard Error of Mean 0.34; effect size: -0.36
Statistical Analysis 4: Comparison: PCIT-Health vs Wait List Control; Difference on difference for number of screens in child bedroom from T3 to T1; Test type: Superiority; p = 0.04, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.91, Standard Error of Mean 0.39; effect size: -0.85

18. Secondary Outcome: Media Parenting Practices (Observed)
Description: Family mealtime observations will be coded for presence and use of screen media (TV, mobile device present, other media present). Coding of the observed behavior is as follows: TV on = 1 if TV is on during mealtime, TV on = 0 if TV is off during mealtime, lower values = better outcomes. Mobile device present = 1 if a mobile device is present, 0 if no mobile device is present, with lower values= better outcomes. Other media present = 1 if other screens are present, 0 if no other screens are present (lower values=better outcomes).
Time Frame: as for outcome 2
Population: Family mealtime recordings were provided by one caregiver.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 11 | 7
score on a scale
  Change in TV on during mealtime from T2 to T1 | -0.39 (0.11) | 0.11 (0.18)
  Change in TV on during mealtime from T3 to T1: number analyzed (Participants) | 8 | 5
  Change in TV on during mealtime from T3 to T1 | -0.33 (0.10) | 0.00 (0.16)
  Change in mobile device present during mealtime from T2 to T1 | -0.09 (0.12) | 0.11 (0.20)
  Change in mobile device present during mealtime from T3 to T1: number analyzed (Participants) | 8 | 5
  Change in mobile device present during mealtime from T3 to T1 | 0.00 (0.11) | 0.29 (0.18)
  Change in other media present during mealtime from T2 to T1 | -0.17 (0.08) | 0.22 (0.13)
  Change in other media present during mealtime from T3 to T1: number analyzed (Participants) | 8 | 5
  Change in other media present during mealtime from T3 to T1 | -0.22 (0.09) | 0.0 (0.14)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for TV on during mealtime from T2 to T1; Test type: Superiority; p = 0.03, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.50, Standard Error of Mean 0.21; effect size: -1.25
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for TV on during mealtime from T3 to T1; Test type: Superiority; p = 0.10, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.33, Standard Error of Mean 0.19; effect size: -1.08
Statistical Analysis 3: Comparison: PCIT-Health vs Wait List Control; Difference on difference for mobile device present during mealtime from T2 to T1; Test type: Superiority; p = 0.41, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.20, Standard Error of Mean 0.24; effect size: -0.44
Statistical Analysis 4: Comparison: PCIT-Health vs Wait List Control; Difference on difference for mobile device present during mealtime from T3 to T1; Test type: Superiority; p = 0.21, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.29, Standard Error of Mean 0.22; effect size: -0.80
Statistical Analysis 5: Comparison: PCIT-Health vs Wait List Control; Difference on difference for other media present during mealtime from T2 to T1; Test type: Superiority; p = 0.02, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.40, Standard Error of Mean 0.16; effect size: -1.29
Statistical Analysis 6: Comparison: PCIT-Health vs Wait List Control; Difference on difference for other media present during mealtime from T3 to T1; Test type: Superiority; p = 0.20, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.22, Standard Error of Mean 0.16; effect size: -0.82

19. Secondary Outcome: Parent Feeding Practices (Observed)
Description: Family mealtime observations will be coded using a modified version of the Mealtime Interaction Coding System. Aspects of task accomplishment (TA) and behavior control BC) were coded. Scores could range from 1 (min) to 3 (max), with higher scores = better outcomes.
Time Frame: as for outcome 2
Population: One caregiver submitted family mealtime observations per family.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 11 | 7
score on a scale
  Change in TA score during mealtime from T2 to T1 | 0.09 (0.07) | -0.33 (0.12)
  Change in TA score during mealtime from T3 to T1: number analyzed (Participants) | 8 | 5
  Change in TA score during mealtime from T3 to T1 | 0.11 (0.08) | 0.14 (0.13)
  Change in BC score during mealtime from T2 to T1 | 0.13 (0.10) | -0.11 (0.17)
  Change in BC score during mealtime from T3 to T1: number analyzed (Participants) | 8 | 5
  Change in BC score during mealtime from T3 to T1 | 0.11 (0.08) | 0.14 (0.13)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for mealtime task accomplishment scores from T2 to T1; Test type: Superiority; p = 0.009, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 0.42, Standard Error of Mean 0.14; effect size: 1.55
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for mealtime task accomplishment scores from T3 to T1; Test type: Superiority; p = 0.84, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.03, Standard Error of Mean 0.15; effect size: -0.13
Statistical Analysis 3: Comparison: PCIT-Health vs Wait List Control; Difference on difference for mealtime behavior control scores from T2 to T1; Test type: Superiority; p = 0.24, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 0.24, Standard Error of Mean 0.20; effect size: 0.63
Statistical Analysis 4: Comparison: PCIT-Health vs Wait List Control; Difference on difference for mealtime behavior control scores from T3 to T1; Test type: Superiority; p = 0.84, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -0.03, Standard Error of Mean 0.15; effect size: -0.13

20. Other Pre Specified Outcome: Child Disruptive Behaviors (Parent Report)
Description: Eyberg Child Behavior Inventory (ECBI); intensity t-score. Higher t-scores indicate poorer outcomes (i.e., greater intensity of behavior problems). T-scores have a mean of 50 (SD = 10). T-scores of 60 or higher indicate clinical significance.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
T-score
  Change in ECBI intensity t-score from T2 to T1 | -8.95 (1.25) | 0.55 (1.77)
  Change in ECBI intensity t-score from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in ECBI intensity t-score from T3 to T1 | -8.74 (1.40) | -1.11 (2.04)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for ECBI intensity t-scores from T2 to T1; Test type: Superiority; p = 0.00, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -9.50, Standard Error of Mean 2.17; effect size: -1.50
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for ECBI intensity t-scores from T3 to T1; Test type: Superiority; p = 0.01, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -7.63, Standard Error of Mean 2.48; effect size: -1.12

21. Other Pre Specified Outcome: Child Psychological Functioning (Parent Report)
Description: Behavior Assessment System for Children (BASC-3); internalizing symptoms t-score (lower scores better outcome) and adaptive skills t-score (higher scores better outcome). T-scores M = 50, SD = 10, with clinical cut-offs at 70 or above.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 21 | 11
T-score
  Change in internalizing symptoms from T2 to T1 | -9.48 (1.54) | -2.55 (2.13)
  Change in internalizing symptoms from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in internalizing symptoms from T3 to T1 | -8.58 (2.02) | -2.00 (2.93)
  Change in adaptive skills from T2 to T1 | -10.2 (4.12) | -3.73 (5.56)
  Change in adaptive skills from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in adaptive skills from T3 to T1 | -13.79 (5.01) | -10.22 (7.27)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for internalizing symptoms from T2 to T1; Test type: Superiority; p = 0.02, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -6.93, Standard Error of Mean 2.63; effect size: -0.93
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for internalizing symptoms from T3 to T1; Test type: Superiority; p = 0.08, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -6.58, Standard Error of Mean 3.56; effect size: -0.68
Statistical Analysis 3: Comparison: PCIT-Health vs Wait List Control; Difference on difference for adaptive skills from T2 to T1; Test type: Superiority; p = 0.36, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = -6.47, Standard Error of Mean 6.92; effect size: -0.33
Statistical Analysis 4: Comparison: PCIT-Health vs Wait List Control; Difference on difference for adaptive skills from T3 to T1; Test type: Superiority; p = 0.69, ANOVA — [p-value comment as in outcome 1, analysis 2]; Repeated measures; Mean Difference (Net) = -3.57, Standard Error of Mean 8.83; effect size: -0.15

22. Other Pre Specified Outcome: Child Psychosocial Strengths (Parent Report)
Description: Psychosocial Strengths Inventory for Children and Adolescents (PSICA). Scores reflect total sum, ranging from 36 (min) to 252 (max); higher scores indicate better outcomes.
Time Frame: as for outcome 2
Population: Note that the n and means/sd reflect multiple caregivers per family. Statistical analysis accounts for nested data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 22 | 11
score on a scale
  Change in PSICA intensity from T2 to T1 | 30.39 (4.16) | -5.39 (5.89)
  Change in PSICA intensity from T3 to T1: number analyzed (Participants) | 19 | 9
  Change in PSICA intensity from T3 to T1 | 28.12 (4.33) | 6.35 (6.29)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference for PSICA intensity scores from T2 to T1 (higher scores indicate better outcomes); Test type: Superiority; p = 0.000, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 35.78, Standard Error of Mean 7.21; effect size: 1.70
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for PSICA intensity scores from T3 to T1; Test type: Superiority; p = 0.01, ANOVA — [p-value comment as in outcome 1, analysis 2]; repeated measures; Mean Difference (Net) = 21.78, Standard Error of Mean 7.64; effect size: 1.04

23. Primary Outcome: Change in Child Body Mass Index (BMI) Z-score
Description: Change in child BMI z-score will be calculated using standardized anthropometric measurement (height and weight) procedure. The z-score is a standard deviation away from the mean, based on the CDC growth charts. Higher z-scores indicate greater weight status. A Z-score of 0 equals the population mean, based on age and sex.
Time Frame: as for outcome 2
Population: For Time 2, n = 11 for PCIT-health and n = 7 for control. For Time 3, n = 9 for PCIT-health and n = 6 for control.
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | PCIT-Health | Wait List Control
Number analyzed (Participants) | 11 | 7
Z-score
  Change in BMI z-score (T2-T1); negative values indicate decrease in BMI z-score | 0.11 (0.08) | 0.06 (0.12)
  Change in BMI z-score (T3-T1); negative values indicate decrease in BMI z-score: number analyzed (Participants) | 9 | 6
  Change in BMI z-score (T3-T1); negative values indicate decrease in BMI z-score | 0.01 (0.10) | 0.02 (0.15)
Statistical Analysis 1: Comparison: PCIT-Health vs Wait List Control; Difference on difference from T2 to T1 for BMI z-score; Test type: Superiority; p = .73, ANOVA — Given this is a pilot RCT, primary aim is to estimate effect size for a more fully-powered RCT. P-values will be provided in addition to effect size; Repeated measures; Mean Difference (Net) = 0.05, Standard Error of Mean 0.14 — Effect size: 0.17
Statistical Analysis 2: Comparison: PCIT-Health vs Wait List Control; Difference on difference for BMI z-scores from T3 to T1; Test type: Superiority; p = .98, ANOVA — [p-value comment as in outcome 23, analysis 1]; Repeated measures; Mean Difference (Net) = 0.00, Standard Error of Mean 0.18; Effect size: -0.01

ADVERSE EVENTS:
Time Frame: During of the study (approximately 10 months)
Description: Weekly check-ins with participants about well-being for families enrolled in the intervention; bimonthly check-ins between baseline and 6 month follow-up for enrolled families. Did not explicitly ask about adverse events, but inquired as to family and child well-being.
Arm/Group | PCIT-Health | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/18
Other Adverse Events (participants affected / at risk) | 0/41 | 0/18

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic necessitated changes to our methodology. We changed our intervention into a telehealth format delivered through synchronous video conferencing and other remote distancing strategies. We had to temporarily suspend in-person data collection for participants in the early part of the pandemic, until distancing guidelines could be adhered to safely with personal protective equipment in our clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03982511/Prot_SAP_002.pdf
  • Informed Consent Form (2019-10-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT03982511/ICF_001.pdf